CLINICAL TRIAL: NCT05590481
Title: Effect of Tibial Transcutaneous Electrostimulation in Women with Urgency Urinary Incontinence Compared to a Sham Group: Randomized Clinical Trial
Brief Title: Effect of Tibial Transcutaneous Electrostimulation in Women with Urgency Urinary Incontinence
Acronym: TibialTNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Leila Katz, Professor Phd Leila Katz, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIBIALTENS
Record Dates: First submitted 2022-08-29; First posted 2022-10-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence, Urge
Keywords: urinary incontinence; Sleep; nocturia; sedentary behavior; anxiety; quality of life
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence; Nocturia; Sedentary Behavior; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EG (experimental group): TIBIAL TRANSCUTANEOUS ELECTROSTIMULATION + Behavioral Therapy (Experimental): EG (experimental group): submitted to a behavioral therapy protocol, which involves bladder training, pelvic floor muscle training and modification of liquid intake. The orientation will be based on the initial evaluation of the patient, in which the responsible researcher will give verbal orientations and deliver booklets on the pathology, behavioral therapy and sleep hygiene. In addition, patients will be submitted to biphasic current and surface electrodes during 12 treatment sessions, twice a week, on non-consecutive days, with a DUALPEX 961s electrical stimulation device (Quark, Brazil).
  Interventions: Device: TIBIAL TRANSCUTANEOUS ELECTROSTIMULATION; Behavioral: behavioral therapy protocol
- GS (Sham-sham group): Behavioral therapy (Sham Comparator): GS (Sham-sham group): submitted to a behavioral therapy protocol, which involves bladder training, pelvic floor muscle training and modification of liquid intake. The orientation will be based on the initial evaluation of the patient, in which the responsible researcher will give verbal orientations and deliver booklets on the pathology, behavioral therapy and sleep hygiene. Twelve sessions will be held, twice a week, on non-consecutive days. The electrodes of the DUALPEX 961 equipment will be positioned one immediately posterior to the lateral malleolus of the ankle and the other approximately 30 cm above it, where there is no stimulus for the tibial nerve.
  Interventions: Behavioral: behavioral therapy protocol

INTERVENTIONS:
Device: TIBIAL TRANSCUTANEOUS ELECTROSTIMULATION — The electrodes will be surface (silicone rubber and carbonate), brand Quark®, with dimensions of 5 cm by 3 cm, coupled with conductive gel and fixed to the volunteer's skin with micropore tape. For the placement of the electrodes, the volunteer will be positioned in the horizontal supine position on the stretcher, with the knee in semiflexion and the head supported on a pillow. The electrodes will be positioned one immediately posterior to the medial malleolus of the ankle and the other approximately 10 cm above it, both fixed with micropore tape, on both legs of the patient. To ensure that the electrodes stimulate the tibial nerve, a transcutaneous electrical nerve stimulation (TENS) current with a frequency of 1 Hz will first be applied, with a gradual increase in intensity, to verify a rhythmic movement of flexion of the hallux. The following parameters will be used for TTNS: frequency 10Hz (Hertz), pulse duration 200 μs (microseconds), for 30 minutes.
  Arms: EG (experimental group): TIBIAL TRANSCUTANEOUS ELECTROSTIMULATION + Behavioral Therapy
Behavioral: behavioral therapy protocol — submitted to a behavioral therapy protocol, which involves bladder training, pelvic floor muscle training and modification of liquid intake. The orientation will be based on the initial evaluation of the patient, in which the responsible researcher will give verbal orientations and deliver booklets on the pathology, behavioral therapy and sleep hygiene.

SUMMARY:
Urge urinary incontinence (UUI) is associated with nocturia, a common cause of sleep disorders, also related to levels of anxiety and depression. Studies demonstrate improvement in the clinical parameters of women with UUI after treatment with transcutaneous tibial nerve stimulation (TTNS). However, there are few data available on the association of urinary symptoms in women with UUI with sedentary behavior (SB), physical activity level (PAL) and sleep quality (SQ). Our study has the objective of evaluating the impact of TTNS on urinary symptoms, anxiety level, life quality(LQ), sleep parameters, PAL and SB in women with UUI.

DETAILED DESCRIPTION:
A randomized clinical trial, sham-controlled, comparing behavioral therapy and TTNS (intervention) to the use of behavioral therapy alone. It will include women with 18 years or more, diagnosed with UUI or mixed IU attested by the Questionnaire Overactive Bladder Validated 8 (OAB-V8).

Women with active urinary tract infection in the last four weeks, alcoholics, smokers or drug addicts, with lesions and alteration of skin sensitivity in the place where electrotherapy will be applied, in drug and/or physiotherapeutic treatment for UUI or current OAB, using sleep-inducing medication, with any neurological disease, using anticholinergic drugs, calcium antagonists, antagonists and dopamine antagonists, with presence of pelvic organ prolapse, during pregnancy or puerperal or with any difficulty in understanding or cognitive deficit that makes it impossible to carry out the research will be excluded.

Study variables are behavioral therapy, bilateral transcutaneous tibial nerve stimulation, type of UI, PAL, excessive daytime sleepiness, generic and specific LQ, SQ, UI severity, anxiety level, urinary frequency, nocturia and bladder capacity.

Sample size was calculated, adopting a two-tailed test with the following parameters: α = 0.05, β = 0.20 and statistical power of 80% and 102 women will be included.

The study will be carried out in two physiotherapy clinics in Recife, from September 2022 to June 2023, both groups will undergo a behavioral therapy protocol, (bladder training, pelvic floor muscle training and modification of liquid intake). Patients will be submitted to biphasic current and surface electrodes during 12 treatment sessions, twice a week, on non-consecutive days, with a electrical stimulation device (Quark, Brazil). The following parameters will be used for TTNS: frequency 10Hz (dez Hertz), pulse duration 200 μs (microseconds), for 30 minutes. In the experimental group, the electrodes will be positioned on the medial malleolus of both legs), in order to stimulate the tibial nerve path. In the Sham group, the electrodes will be placed on both legs, centered in the middle of the thigh, where there is no stimulus for the tibial or sacral nerve, for 30 minutes.

The project was approved by the Research Ethics Committee of Professor Fernando Figueira Institute of Integral Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Age from 18 years old;
* Diagnosis of urgency urinary incontinence or mixed urinary incontinence
* Score greater than or equal to 8 on the Hyperactive Bladder - Validated 8 Question Awareness Tool (OAB-V8)

Exclusion Criteria:

* -Active urinary infection in the last four weeks;
* Alcoholism, smoking or drug addiction;
* Lesions and alteration of skin sensitivity in the place where electrotherapy will be applied;
* Drug and/or physiotherapeutic treatment for urgency urinary incontinence;
* Use of sleep-inducing medication,
* Any neurological disease (multiple sclerosis, Alzheimer's disease, stroke and Parkinson's disease);
* Use of anticholinergic drugs, calcium antagonists, b-antagonists and dopamine antagonists;
* Presence of pelvic organ prolapse (POP), measured by a score greater than III by the POP-Q system;
* Any comprehension difficulty or cognitive deficit that makes it impossible to carry out the research;
* Gestational or puerperal period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Nocturia | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  People with an overactive bladder can experience nocturia, which means they need to get up frequently at night to go to the bathroom. Nocturia will be evaluated through the voiding diary that the volunteers will be instructed to complete. The more times the volunteer gets up at night to urinate, the more severe the condition.

SECONDARY OUTCOMES:
sleep quality | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Assessed by the Pittsburgh Sleep Quality Index (PSQI), with the global score ranging from 0 to 21. The higher, the worse the sleep quality.
physical activity level | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  lifestyle based on the daily number of steps
sedentary behavior | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  lifestyle based on the daily number of steps
anxiety level | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  A mental health disorder characterized by feelings of worry, anxiety, or fear that are strong enough to interfere with daily activities. Screening for study anxiety will be performed using the the Hospital Anxiety and Depression Scale (HADS). The scale is validated for Portuguese and was developed to identify possible cases of anxiety and depression through a structured and easy-to-apply questionnaire.The HADS consists of two subscales of 14 varied questions: 7 questions that measure anxiety (HADS-A) and 7 that measure depression (HADS-D). Each question has four possible answers and a score from 0 to 3 is given. The total score is then calculated and can range between 0 and 21 points on each subscale, with a higher score indicating more severe symptoms. The cut-off score for "possible cases" of anxiety and depression is 8 points or higher, which is the cut-off identified to provide the optimal balance between specificity and sensitivity.
Sleep parameters - Total time of sleep | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Total time the individual spent sleeping during the night
Excessive daytime sleepiness | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  discrete quantitative variable, assessed using the Epworth sleepiness scale 1 ( ) yes, 2 ( ) no. It is a self-administered questionnaire and refers to the possibility of napping in eight everyday situations.
Severity of urinary incontinence | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  To identify how much the urinary incontinence impacts one's life.The severity of UI will be assessed using the Incontinence Severity Index (ISI), translated and validated into Portuguese by Pereira et al, in 2011 (Appendix 1)(126). This instrument consists of two questions regarding the frequency (1-4 points) and amount (1-3 points) of urinary loss. To obtain the final score, the scores for frequency of urinary leakage and the amount of urinary leakage are multiplied.
Life's quality | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  The SF-36 Medical Outcomes Study 36 - Item Short - Form Health Survey (SF36) is a generic instrument for assessing quality of life that is easy to administer and understand. It consists of a multidimensional questionnaire, consisting of 36 items, encompassed in 8 scales or domains. It has a final score from 0 to 100 (obtained by calculating the Raw Scale), where 0 corresponds to the worst general health status and 100 corresponds to the best health status.
Sleep parameters - sleep efficiency | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Sleep efficiency is the relationship between the time the patient spent in bed and the actual sleep time.
Sleep parameters - Total time in bed | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Total time in bed, whether sleeping or not.
Sleep parameters - Nightly awakenings | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Number of times the individual wakes up during the night
Sleep parameters - Time awake after falling asleep | Baseline/ change after the 6th week of treatment /change 30 days after the 6th week of treatment(follow up).
  Time awake after sleep started, total time of nocturnal awakenings.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Katz, PHD, Principal Investigator — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Instituto de medicina integral fernando figueira, Recife, Pernambuco, Brazil